CLINICAL TRIAL: NCT01291108
Title: Safety and Efficacy of AGN-210669 Ophthalmic Solution Compared With Bimatoprost Ophthalmic Solution in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210669-013
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Results first posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- AGN-210669 (Experimental): AGN-210669 0.05% applied as 1 drop in both eyes every evening during Month 1.
  Interventions: Drug: AGN-210669
- AGN-210669 + bimatoprost (Experimental): AGN-210669 0.05% + bimatoprost ophthalmic solution 0.03% applied as 1 drop of each treatment in both eyes every evening during Month 2.
  Interventions: Drug: AGN-210669; Drug: bimatoprost
- AGN-210669 + bimatoprost vehicle (Experimental): AGN-210669 0.05% + bimatoprost ophthalmic solution 0.03% vehicle applied as 1 drop of each treatment in both eyes every evening during Month 2.
  Interventions: Drug: AGN-210669; Drug: bimatoprost vehicle
- bimatoprost (Active Comparator): bimatoprost ophthalmic solution 0.03% applied as 1 drop in both eyes every evening during Month 1.
  Interventions: Drug: bimatoprost
- bimatoprost + AGN-210669 (Experimental): bimatoprost ophthalmic solution 0.03% + AGN-210669 0.05% applied as 1 drop of each treatment in both eyes every evening during Month 2.
  Interventions: Drug: AGN-210669; Drug: bimatoprost
- bimatoprost + bimatoprost vehicle (Other): bimatoprost ophthalmic solution 0.03% + bimatoprost ophthalmic solution 0.03% vehicle applied as 1 drop of each treatment in both eyes every evening during Month 2.
  Interventions: Drug: bimatoprost; Drug: bimatoprost vehicle

INTERVENTIONS:
Drug: AGN-210669 — AGN-210669 0.05% applied as 1 drop in both eyes every evening during Month 1 or Month 2.
  Arms: AGN-210669; AGN-210669 + bimatoprost; AGN-210669 + bimatoprost vehicle; bimatoprost + AGN-210669
Drug: bimatoprost — bimatoprost ophthalmic solution 0.03% applied as 1 drop in both eyes every evening during Month 1 or Month 2.
  Other Names: LUMIGAN®
  Arms: AGN-210669 + bimatoprost; bimatoprost; bimatoprost + AGN-210669; bimatoprost + bimatoprost vehicle
Drug: bimatoprost vehicle — bimatoprost ophthalmic solution 0.03% vehicle applied as 1 drop in both eyes every evening during Month 2.
  Arms: AGN-210669 + bimatoprost vehicle; bimatoprost + bimatoprost vehicle

SUMMARY:
This study will evaluate the safety and efficacy of AGN-210669 ophthalmic solution compared with bimatoprost ophthalmic solution (Lumigan®) as monotherapy and adjunctive therapy in patients with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma or ocular hypertension in each eye
* Requires bilateral treatment with an IOP-lowering medication
* Best corrected visual acuity of 20/100 or better in each eye

Exclusion Criteria:

* Use of oral, intramuscular, intravenous or topical ophthalmic corticosteroids within 2 months
* Inability to fast for up to 10 hours
* Prior refractive laser surgery (eg, LASIK, radial keratectomy, photorefractive keratectomy)
* Intraocular surgery or IOP-lowering laser surgery (eg, laser trabeculoplasty) within 6 months
* Current or anticipated use of artificial tears or any ocular medications aside from study medications during study
* Anticipated wearing of contact lenses during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pts were randomized at Baseline for the entire study. At Mo 1, pts received either AGN-210669 or bimatoprost. At Mo 2, pts who had received AGN-210669, then received either AGN-210669+bimatoprost or AGN-210669+bimatoprost vehicle and pts who had received bimatoprost, then received either bimatoprost+AGN-210669 or bimatoprost+bimatoprost vehicle.
Period: Month 1 (Monotherapy)
Arm/Group | AGN-210669 | AGN-210669 + Bimatoprost | AGN-210669 + Bimatoprost Vehicle | Bimatoprost | Bimatoprost + AGN-210669 | Bimatoprost + Bimatoprost Vehicle
Started | 65 | 0 | 0 | 60 | 0 | 0
Completed | 64 (All patients who completed Month 1 were randomized to adjunctive therapy for Month 2.) | 0 | 0 | 60 (All patients who completed Month 1 were randomized to adjunctive therapy for Month 2.) | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Period: Month 2 (Adjunctive Therapy)
Arm/Group | AGN-210669 | AGN-210669 + Bimatoprost | AGN-210669 + Bimatoprost Vehicle | Bimatoprost | Bimatoprost + AGN-210669 | Bimatoprost + Bimatoprost Vehicle
Started | 0 (All patients who completed Month 1 were randomized to adjunctive therapy for Month 2.) | 40 | 24 | 0 (All patients who completed Month 1 were randomized to adjunctive therapy for Month 2.) | 34 | 26
Completed | 0 | 38 | 24 | 0 | 34 | 25
Not Completed | 0 | 2 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- AGN-210669 Followed by AGN-210669 + Bimatoprost: AGN-210669 0.05% applied as 1 drop in each eye every evening for Month 1 followed by AGN-210669 0.05% + bimatoprost 0.03% applied as 1 drop of each treatment in both eyes every evening for Month 2.
- AGN-210669 Followed by AGN-210669 + Bimatoprost Vehicle: AGN-210669 0.05% applied as 1 drop in each eye every evening for Month 1 followed by AGN-210669 0.05% + bimatoprost 0.03% vehicle applied as 1 drop of each treatment in both eyes every evening for Month 2.
- Bimatoprost Followed by Bimatoprost + AGN-210669: bimatoprost 0.03% applied as 1 drop in each eye every evening for Month 1 followed by bimatoprost 0.03% + AGN-210669 applied as 1 drop of each treatment in both eyes every evening for Month 2.
- Bimatoprost Followed by Bimatoprost + Bimatoprost Vehicle: bimatoprost 0.03% applied as 1 drop in each eye every evening for Month 1 followed by bimatoprost 0.03% + bimatoprost 0.03% vehicle applied as 1 drop of each treatment in both eyes every evening for Month 2.
- Total: Total of all reporting groups
Arm/Group | AGN-210669 Followed by AGN-210669 + Bimatoprost | AGN-210669 Followed by AGN-210669 + Bimatoprost Vehicle | Bimatoprost Followed by Bimatoprost + AGN-210669 | Bimatoprost Followed by Bimatoprost + Bimatoprost Vehicle | Total
Number analyzed (Participants) | 44 | 21 | 40 | 20 | 125
Age, Customized [Number; unit: Participants]
  <45 years | 1 | 1 | 1 | 0 | 3
  45 to 65 years | 17 | 10 | 20 | 7 | 54
  >65 years | 26 | 10 | 19 | 13 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 15 | 27 | 13 | 82
  Male | 17 | 6 | 13 | 7 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Eye IOP
Description: IOP is a measurement of the fluid pressure inside the eye. The average of the 2 eyes are used for the analyses. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening). Data are recorded at Hours 0, 4, 8, and 12.
Time Frame: Baseline, Day 57
Population: Modified Intent to Treat: all randomized and treated patients who had a baseline and at least 1 post-baseline IOP measurement
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Groups:
- AGN-210669 Followed by AGN-210669 + Bimatoprost Vehicle: AGN-210669 0.05% + bimatoprost ophthalmic solution 0.03% vehicle applied as 1 drop of each treatment in both eyes every evening during Month 2.
- Bimatoprost Followed by Bimatoprost + Bimatoprost Vehicle: bimatoprost ophthalmic solution 0.03% + bimatoprost ophthalmic solution 0.03% vehicle applied as 1 drop of each treatment in both eyes every evening during Month 2.
- Combined Adjunctives: Combined adjunctives refer to the combined groups of 'AGN-210669 0.05% + bimatoprost' and 'bimatoprost + AGN-210669 0.05%'. The first treatment is applied as 1 drop in each eye every evening for Month 1 followed by AGN-210669 0.05% + bimatoprost 0.03% applied as 1 drop of each treatment in both eyes every evening for Month 2.
Arm/Group | AGN-210669 Followed by AGN-210669 + Bimatoprost Vehicle | Bimatoprost Followed by Bimatoprost + Bimatoprost Vehicle | Combined Adjunctives
Number analyzed (Participants) | 24 | 26 | 75
Millimeters of Mercury (mmHg)
  Baseline - Hour 0 | 26.16 (2.169) | 25.98 (1.962) | 26.26 (2.446)
  Baseline - Hour 4 | 23.91 (2.382) | 23.82 (2.301) | 23.85 (2.553)
  Baseline - Hour 8 | 22.49 (1.338) | 22.35 (2.024) | 22.79 (2.391)
  Baseline - Hour 12 | 21.48 (2.467) | 22.07 (2.596) | 21.73 (2.624)
  Change from Baseline at Day 57-Hr 0 (n=24,25,72) | -7.57 (2.881) | -10.28 (3.190) | -10.84 (3.460)
  Change from Baseline at Day 57-Hr 4 (n=24,25,72) | -6.95 (2.503) | -8.95 (3.531) | -8.79 (3.330)
  Change from Baseline at Day 57-Hr 8 (n=24,25,72) | -5.57 (3.484) | -7.19 (3.198) | -7.67 (2.596)
  Change from Baseline at Day 57-Hr 12 (n=16,17,56) | -5.31 (2.690) | -6.87 (2.838) | -6.03 (2.642)

2. Secondary Outcome: Change From Baseline in Worse Eye IOP
Description: IOP is a measurement of the fluid pressure inside the eye. The worse eye IOP refers to eye with the worse baseline IOP, which is determined as the eye with the higher mean diurnal IOP at baseline. If both eyes have the same mean diurnal IOP at baseline, the right eye is designated as the worse eye. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening). Data are recorded at Hours 0, 4, 8, and 12.
Time Frame: Baseline, Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | AGN-210669 Followed by AGN-210669 + Bimatoprost Vehicle | Bimatoprost Followed by Bimatoprost + Bimatoprost Vehicle | Combined Adjunctives
Number analyzed (Participants) | 24 | 26 | 75
Millimeters of Mercury (mmHg)
  Baseline - Hour 0 | 26.56 (2.305) | 26.40 (2.069) | 26.61 (2.664)
  Baseline - Hour 4 | 24.60 (2.754) | 24.25 (2.295) | 24.31 (2.685)
  Baseline - Hour 8 | 23.04 (1.687) | 22.73 (2.290) | 23.17 (2.591)
  Baseline - Hour 12 | 21.72 (2.811) | 22.47 (2.598) | 21.93 (2.908)
  Change from Baseline at Day 57-Hr 0 (n=24,25,72) | -7.50 (2.989) | -10.56 (3.435) | -10.96 (3.705)
  Change from Baseline at Day 57-Hr 4 (n=24,25,72) | -7.38 (2.841) | -9.16 (3.472) | -9.01 (3.515)
  Change from Baseline at Day 57-Hr 8 (n=24,25,72) | -5.94 (3.817) | -7.42 (3.526) | -7.92 (3.002)
  Change from Baseline at Day 57-Hr 12 (n=16,17,56) | -5.00 (2.696) | -7.00 (2.969) | -5.99 (3.076)

ADVERSE EVENTS:
Description: The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs) and included all treated patients. SAEs and AEs are presented by treatment arm not necessarily by individual treatment received.
Arm/Group | AGN-210669 | AGN-210669 + Bimatoprost | AGN-210669 + Bimatoprost Vehicle | Bimatoprost | Bimatoprost + AGN-210669 | Bimatoprost + Bimatoprost Vehicle
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/40 | 0/24 | 0/60 | 0/34 | 1/26
Other Adverse Events (participants affected / at risk) | 43/65 | 31/40 | 11/24 | 41/60 | 26/34 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-210669 (N=65) | AGN-210669 + Bimatoprost (N=40) | AGN-210669 + Bimatoprost Vehicle (N=24) | Bimatoprost (N=60) | Bimatoprost + AGN-210669 (N=34) | Bimatoprost + Bimatoprost Vehicle (N=26)
Uveal Prolapse (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-210669 (N=65) | AGN-210669 + Bimatoprost (N=40) | AGN-210669 + Bimatoprost Vehicle (N=24) | Bimatoprost (N=60) | Bimatoprost + AGN-210669 (N=34) | Bimatoprost + Bimatoprost Vehicle (N=26)
Corneal Thickening (Eye disorders) | 19 | 10 | 4 | 2 | 15 | 0
Conjunctival Hyperaemia (Eye disorders) | 17 | 23 | 2 | 24 | 13 | 5
Eye Irritation (Eye disorders) | 6 | 4 | 1 | 2 | 3 | 1
Eye Discharge (Eye disorders) | 5 | 3 | 0 | 3 | 1 | 1
Vision Blurred (Eye disorders) | 5 | 5 | 0 | 3 | 5 | 0
Eye Pruritus (Eye disorders) | 4 | 3 | 0 | 4 | 5 | 0
Punctate Keratitis (Eye disorders) | 3 | 6 | 3 | 7 | 4 | 4
Photophobia (Eye disorders) | 3 | 10 | 0 | 4 | 12 | 1
Foreign Body Sensation in Eyes (Eye disorders) | 2 | 5 | 0 | 6 | 3 | 0
Eye Pain (Eye disorders) | 0 | 9 | 1 | 0 | 8 | 2
Lacrimation Increased (Eye disorders) | 3 | 2 | 0 | 0 | 2 | 0
Iritis (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0
Anterior Chamber Cell (Eye disorders) | 0 | 2 | 0 | 0 | 1 | 2
Asthenopia (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.